CLINICAL TRIAL: NCT03079765
Title: Training Educators to Implement Behavioral Assessment and Treatment Procedures in School Settings Via Telehealth
Brief Title: Training Educators to Conduct Functional Behavior Assessment Via Telehealth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 16-1691
Record Dates: First submitted 2017-03-08; First posted 2017-03-14 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Autism Spectrum Disorder
Keywords: Telehealth; Functional behavior assessment
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline (Experimental): Participants will be given a written protocol for conducting the relevant assessment procedure (e.g., open-ended interview).
  Interventions: Behavioral: Protocol Only
- Telehealth Treatment (Active Comparator): Participants will receive feedback and error correction on their implementation of the relevant assessment procedure to improve their performance.
  Interventions: Behavioral: Behavioral skills training; Behavioral: Protocol Only

INTERVENTIONS:
Behavioral: Behavioral skills training — Participants will receive feedback and error correction on their implementation of the assessment procedures. Feedback will take the form of the experimenter pointing out components of the assessment that are not being conducted accurately and error correction will take the form of the experimenter reviewing the correct way to implement that component of the assessment.
  Arms: Telehealth Treatment
Behavioral: Protocol Only — Participants will be given a written protocol describing how to conduct the target assessment procedure.

SUMMARY:
This study evaluates the effects of delivering training services via telehealth to educators in rural schools. The investigators hope to increase the accuracy with which educators implement functional behavior assessments in schools. During the study, participants will receive training on functional behavior assessments at different periods. When one school is receiving training, other schools will not be receiving training. The purpose will be to show increased accuracy of functional behavior assessments only occur following training.

DETAILED DESCRIPTION:
Training services for educators typically occurs in-vivo with experts providing immediate feedback and modeling to shape behavior. These types of training experiences may not be accessible for all educators though. The current study will evaluate delivering behavioral skills training (e.g., feedback and error correction) via telehealth for educators conducting functional behavior assessments. The components of the functional behavior assessment that will be targeted are open-ended interviews, stimulus preference assessments, direct observations of problem behavior, and a functional communication training program. With at least three different schools, the investigators will introduce training delivered via telehealth one at a time to show that increases in acquisition of the various components of the functional behavior assessment only occur following telehealth-based training.

ELIGIBILITY:
Inclusion Criteria:

* Must be an educator who conducts functional behavior assessment.
* Must be training to become a registered behavior technician.

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Increased functional behavior assessment procedural fidelity | 1 hour
  Will measure percentage of components of each assessment correctly implemented.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Romani, Ph.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will only be disseminated via professional meetings and peer-reviewed publications. Data will be de-identified to maintain confidentiality of participants. Data will not be shared with anyone else.